CLINICAL TRIAL: NCT03313583
Title: French Transfusion Recipients Cross Sectional Study : Get to Know the Transfusion Recipients Population
Brief Title: French One Day Survey in 2011 - Knowing Our Population of Labile Blood Products Recipients
Acronym: PopReceveur
Status: Completed | Type: Observational
Sponsor: Etablissement Français du Sang (Other)
Collaborators: Centre Hospitalier Universitaire de Besancon (Other); Centre Hospitalier Universitaire de Nice (Other); Assistance Publique Hopitaux De Marseille (Other); Région Nord-Pas de Calais, France (Other)
Responsible Party: Sponsor
Other Study IDs: EFS/2011/PopReceveur
Record Dates: First submitted 2017-09-29; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Blood Product Transfusion for All Conditions; Trauma; Surgical Blood Loss; Hematologic Diseases
MeSH Terms: conditions — Wounds and Injuries; Blood Loss, Surgical; Hematologic Diseases | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood product recipients: All patients who received at least one blood product on the day of the study
  Interventions: Procedure: Transfusion of blood products

INTERVENTIONS:
Procedure: Transfusion of blood products

SUMMARY:
Describe the epidemiologic profile and clinical context of transfusion recipients in France. Describe the clinical context of transfusion.

Describe the characteristics of the transfusion prescriptions, the use of blood products and the main indications for transfusion.

Describe transfusion practice according the type of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

• Transfusion with at least one blood product on the day of the study.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All blood products recipients
Study Population: french population of recipients
Sampling Method: Probability Sample
Enrollment: 4720 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2011-11-01 (Actual); Study Completion 2011-12-01 (Actual)

PRIMARY OUTCOMES:
Number of red blood cell concentrates received | 1 day (cross sectional)
  transversal study
Number of platelet concentrates recevied | 1 day (cross sectional)
  transversal study
Number of plasma units received | 1 day (cross sectional)
  transversal study

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fillet AM, Desmarets M, Assari S, Quaranta JF, Francois A, Pugin A, Schuhmacher A, Lassale B, Monnet E, Cabre P, Legrand D, Binda D, Djoudi R. Blood products use in France: a nationwide cross-sectional survey. Transfusion. 2016 Dec;56(12):3033-3041. doi: 10.1111/trf.13887. Epub 2016 Nov 2. PMID 27807857